CLINICAL TRIAL: NCT05800002
Title: Intravascular Ultrasound Versus Angiography Guided Drug-eluting Stent Implantation for Patients With Coronary Severe Calcification: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: IVUS-guided DES Implantation in Coronary Calcification
Acronym: ULTIMATE IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Junjie Zhang, Vice chief, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20230310-10
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional; Cerebral Angiography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular ultrasound guidance (Experimental)
  Interventions: Procedure: Intravascular ultrasound
- Angiography guidance (Active Comparator)
  Interventions: Procedure: Angiography

INTERVENTIONS:
Procedure: Intravascular ultrasound — Pretreatment strategy, stent size, stent landing zone and post-dilation balloon size are depended on intravascular ultrasound.
  Arms: Intravascular ultrasound guidance
Procedure: Angiography — Pretreatment strategy, stent size, stent landing zone and post-dilation balloon size are depended on angiography.
  Arms: Angiography guidance

SUMMARY:
Coronary calcified lesion is associated with a poor clinical outcome. Intravascular ultrasound (IVUS) provides anatomic information in detail about reference vessel dimensions and lesion characteristics including severity of diameter stenosis, lesion length, and morphology. Both randomized and observational studies have reported the clinical benefits of IVUS guidance for patients with chronic total occlusion (CTO), long lesions, acute coronary syndrome (ACS) with complex bifurcation lesions. Our previous ULTIMATE trial has demonstrated that IVUS-guided drug-eluting stent (DES) implantation significantly improved clinical outcome in all-comers, particularly for patients who had an IVUS-defined optimal procedure, compared with angiography guidance. However, the benefit of IVUS guidance in coronary severe calcification still remains unknown in the modern DES era.

ELIGIBILITY:
Inclusion Criteria:

1. Silent ischemia, stable or unstable angina, non-ST-segment elevation myocardial infarction > 48 hours, or ST-segment elevation myocardial infarction > 7 days;
2. De novo coronary lesion eligible for drug-eluting stent implantation;
3. Target lesion with severe calcification;

Exclusion Criteria:

1. Age less than 18-year-old;
2. Comorbidity with a life expectancy <12 months;
3. Intolerant of antithrombotic therapy;
4. Significant anemia, thrombocytopenia, or leucopenia;
5. History of major hemorrhage (intracranial, gastrointestinal, and so on);
6. Chronic total occlusion lesion not recanalized;
7. Scheduled major surgery in the next 12 months;
8. Left ventricular ejection fraction < 25%;
9. Uremia dependent on dialysis treatment;
10. Previous drug-eluting stent implantation in target vessel;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2033-03-30 (Estimated)

PRIMARY OUTCOMES:
the rate of target-vessel failure at 12 months | 12 months after indexed procedure
  the composite of cardiovascular death, target-vessel myocardial infarction, and clinically driven target-vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided